CLINICAL TRIAL: NCT04744987
Title: Changes in Serum Creatinine Levels Can Help Distinguish Hypovolemic From Euvolemic Hyponatremia
Status: Completed | Type: Observational
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Jorge Gabriel Ruiz Sánchez, Principal investigator, Hospital San Carlos, Madrid
Other Study IDs: creatinine-hyponatremia
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Hyponatremia; Hypovolemia; SIADH
Keywords: hyponatremia diagnosis; serum creatinine;; hypovolemic hyponatremia; euvolemic hyponatremia; SIAD
MeSH Terms: conditions — Hyponatremia; Hypovolemia; Inappropriate ADH Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypovolemic hyponatremia: Patients with any cause of hypovolemic hyponatremia were included.
- Euvolemic hyponatremia: Only patients with euvolemic hyponatremia secondary to Syndrome of inappropriate antidiuresis were included.

SUMMARY:
Retrospective study that analyzes the changes in serum creatinine as a tool to correctly classify the volemic status volemic status (euvolemia vs hypovolemia) of the patients with hyponatremia.

DETAILED DESCRIPTION:
This study evaluates the usefulness of the changes in serum creatinine in differentiating between euvolemia and hypovolemia in hyponatremic patients. Changes in serum creatinine were retrospectively analyzed . The latter was calculated subtracting the serum creatinine value of eunatremia from that of hyponatremia, and was categorized as an increase when it was "positive", or "decrease/no change" when it was negative or equal to zero. The percentual change in serum creatinine was also calculated.

Two groups of patients were selected for the current study. First group was conformed by patients with hypovolemic hyponatremia, and second group by patients with euvolemic hyponatremia. Data from eunatremia as well as the hyponatremic episode were collected. Both groups were matched in Receiver operating characteristic curve analyzes where both arithmetical and percentual changes in serum creatinine were assessed and cut-off points were selected for an additional Odd Ratio analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypovolemic hyponatremia secondary to any cause
* Patients with euvolemic hyponatremia caused by Syndrome of inappropriate antidiuresis
* Complete clinical volemia assessment during hyponatremia.
* Presence of serum creatinine measured in eunatremia as well as in hyponatremic episodes.

Exclusion Criteria:

* Pregnants.
* Patients with a prior history of diabetes, advanced chronic kidney disease (glomerular filtrate rate below 30 ml/min), cirrhosis, or heart failure were excluded.
* Patients with hypervolemic hyponatremia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting with hyponatremia, followed in the monographic Hyponatremia outpatient clinic of the Endocrinology and Nutrition Department of the Hospital Clínico San Carlos, Madrid, Spain. Patients were attended from January 1st 2014 through November 30th 2019.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy of the changes in serum creatinine for volemic classification of hyponatremia | 4 months
  Area under the curve from the Receiver operating characteristic curve analysis were calculated for the changes in serum creatinine. Probabilities of each evaluated tool (arithmetic and percentual change in serum creatinine) to correctly classified the volemic status of the hyponatremic patients were calculated.

SECONDARY OUTCOMES:
Ratio of Correct volemic classification of hyponatremia when Changes in Serum creatinine were used. | 4 months
  Ratio of patients who were correctly classified according to volemic status with different cut-off points obtained from the Receiver operating characteristic curve analyzes. Sensitivity, Specificity, Positive and Negative predictive values were also calculated.
Diagnostic Accuracy of Urine sodium for volemic classification of hyponatremia | 4 months
  Area under the curve from the Receiver operating characteristic curve analysis were calculated for the urine sodium y patients with hyponatremia. Sensitivity, specificity, and Positive and Negative predictive values were calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Runkle, MDPhD, Study Director — Hospital San Carlos, Madrid; Jorge G Ruiz, MD, Principal Investigator — Hospital San Carlos, Madrid
Locations (1):
- Servicio de Endocrinología y Nutrición. Hospital Clínico San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
The data supporting the findings of this study will be available to be requested to the investigators.
Time Frame: starting 12 months after publication to 18 months after publication
Access Criteria: IPD might be requested only by e-mail. IPD might be shared only with medical investigators with a corroborated affiliation and attached to an official research group. IPD would be shared only for an exploratory analysis in order to confirm the results of the current study. IPD sharing request must include reasons for the petition. No new results, research, or publications can be made with the shared IPD. IPD sharing requests will be reviewed and approved by all authors to decide whether to submit.

REFERENCES:
- [Background] Spasovski G, Vanholder R, Allolio B, Annane D, Ball S, Bichet D, Decaux G, Fenske W, Hoorn EJ, Ichai C, Joannidis M, Soupart A, Zietse R, Haller M, van der Veer S, Van Biesen W, Nagler E; Hyponatraemia Guideline Development Group. Clinical practice guideline on diagnosis and treatment of hyponatraemia. Eur J Endocrinol. 2014 Feb 25;170(3):G1-47. doi: 10.1530/EJE-13-1020. Print 2014 Mar. PMID 24569125
- [Background] Verbalis JG, Goldsmith SR, Greenberg A, Korzelius C, Schrier RW, Sterns RH, Thompson CJ. Diagnosis, evaluation, and treatment of hyponatremia: expert panel recommendations. Am J Med. 2013 Oct;126(10 Suppl 1):S1-42. doi: 10.1016/j.amjmed.2013.07.006. PMID 24074529
- [Background] Adrogue HJ, Madias NE. Hyponatremia. N Engl J Med. 2000 May 25;342(21):1581-9. doi: 10.1056/NEJM200005253422107. No abstract available. PMID 10824078
- [Background] Chung HM, Kluge R, Schrier RW, Anderson RJ. Clinical assessment of extracellular fluid volume in hyponatremia. Am J Med. 1987 Nov;83(5):905-8. doi: 10.1016/0002-9343(87)90649-8. PMID 3674097
- [Background] Musch W, Thimpont J, Vandervelde D, Verhaeverbeke I, Berghmans T, Decaux G. Combined fractional excretion of sodium and urea better predicts response to saline in hyponatremia than do usual clinical and biochemical parameters. Am J Med. 1995 Oct;99(4):348-55. doi: 10.1016/s0002-9343(99)80180-6. PMID 7573088
- [Background] Fenske W, Stork S, Koschker AC, Blechschmidt A, Lorenz D, Wortmann S, Allolio B. Value of fractional uric acid excretion in differential diagnosis of hyponatremic patients on diuretics. J Clin Endocrinol Metab. 2008 Aug;93(8):2991-7. doi: 10.1210/jc.2008-0330. Epub 2008 May 13. PMID 18477658
- [Background] Musch W, Decaux G. Utility and limitations of biochemical parameters in the evaluation of hyponatremia in the elderly. Int Urol Nephrol. 2001;32(3):475-93. doi: 10.1023/a:1017586004688. PMID 11583374
- [Background] Musch W, Decaux G. Treating the syndrome of inappropriate ADH secretion with isotonic saline. QJM. 1998 Nov;91(11):749-53. doi: 10.1093/qjmed/91.11.749. PMID 10024938
- [Background] Tzoulis P, Runkle-De la Vega I. The Diagnostic Approach to the Patient with Hyponatremia: Are the Correct Investigations Being Done? Front Horm Res. 2019;52:190-199. doi: 10.1159/000493248. Epub 2019 Jan 15. PMID 32097921
- [Background] Cui H, He G, Yang S, Lv Y, Jiang Z, Gang X, Wang G. Inappropriate Antidiuretic Hormone Secretion and Cerebral Salt-Wasting Syndromes in Neurological Patients. Front Neurosci. 2019 Nov 8;13:1170. doi: 10.3389/fnins.2019.01170. eCollection 2019. PMID 31780881
- [Background] Narins RG, Jones ER, Stom MC, Rudnick MR, Bastl CP. Diagnostic strategies in disorders of fluid, electrolyte and acid-base homeostasis. Am J Med. 1982 Mar;72(3):496-520. doi: 10.1016/0002-9343(82)90521-6. PMID 7036739
- [Background] Cook DJ, Simel DL. The Rational Clinical Examination. Does this patient have abnormal central venous pressure? JAMA. 1996 Feb 28;275(8):630-4. No abstract available. PMID 8594245
- [Background] Avcil M, Kapci M, Dagli B, Omurlu IK, Ozluer E, Karaman K, Yilmaz A, Zencir C. Comparision of ultrasound-based methods of jugular vein and inferior vena cava for estimating central venous pressure. Int J Clin Exp Med. 2015 Jul 15;8(7):10586-94. eCollection 2015. PMID 26379848
- [Background] Nik Muhamad NA, Safferi RS, Robertson CE. Internal Jugular Vein Height and Inferior Vena Cava Diameter Measurement using Ultrasound to Determine Central Venous Pressure: A Correlation Study. Med J Malaysia. 2015 Apr;70(2):63-6. PMID 26162379
- [Background] Rizkallah J, Jack M, Saeed M, Shafer LA, Vo M, Tam J. Non-invasive bedside assessment of central venous pressure: scanning into the future. PLoS One. 2014 Oct 3;9(10):e109215. doi: 10.1371/journal.pone.0109215. eCollection 2014. PMID 25279995
- [Background] Ruiz-Sanchez JG, Meneses D, Alvarez-Escola C, Cuesta M, Calle-Pascual AL, Runkle I. The Effect of the Dose of Isotonic Saline on the Correction of Serum Sodium in the Treatment of Hypovolemic Hyponatremia. J Clin Med. 2020 Nov 5;9(11):3567. doi: 10.3390/jcm9113567. PMID 33167557
- [Background] Soni SS, Adikey GK, Raman AS. Fractional excretion of uric acid as a therapeutic monitor in cerebral salt wasting syndrome. Saudi J Kidney Dis Transpl. 2008 Jan;19(1):106-8. No abstract available. PMID 18087137
- [Background] Oh JY, Shin JI. Syndrome of inappropriate antidiuretic hormone secretion and cerebral/renal salt wasting syndrome: similarities and differences. Front Pediatr. 2015 Jan 22;2:146. doi: 10.3389/fped.2014.00146. eCollection 2014. PMID 25657991
- [Background] Imbriano LJ, Mattana J, Drakakis J, Maesaka JK. Identifying Different Causes of Hyponatremia With Fractional Excretion of Uric Acid. Am J Med Sci. 2016 Oct;352(4):385-390. doi: 10.1016/j.amjms.2016.05.035. Epub 2016 Jul 6. PMID 27776720